CLINICAL TRIAL: NCT00849615
Title: A Prospective Multicenter Study With 5-FU, Leucovorin, Oxaliplatin and Docetaxel (FLOT) in Patients With Locally Advanced, Limited Metastatic or Extensive Metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Brief Title: Prospective Study With FLOT in Patients With Locally Advanced, Limited Metastatic or Extensive Metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Acronym: FLOT3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S396 FLOT3
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Cancer; Adenocarcinoma of the Esophagogastric Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLOT (Experimental)
  Interventions: Drug: Docetaxel; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: folinic acid

INTERVENTIONS:
Drug: Docetaxel — 50mg/m2 qd15
Drug: 5-Fluorouracil — 2600mg/m2 qd15
Drug: Oxaliplatin — 85mg/m2 qd15
Drug: folinic acid — 200mg/m2 qd15

SUMMARY:
Patients with locally advanced or metastatic gastric carcinoma or carcinoma of the esophagogastric junction without prior palliative therapy will be treated with 8 cycles of the FLOT scheme (up to 12 cycles if the response is favourable). Prior to enrollment a unique and detailed clinical evaluation of the dissemination of the disease will be done which includes a differentiated regard of the metastatic status. patients will be classified as having either (A) locally advanced, (B) limited metastatic, or (C) extensive metastatic disease. In arms A and B surgical intervention is planned if operability is reached. The hypothesis is that by classifying patients more individually by the state of their disease, patients in arm B will have a significantly prolonged overall survival compared to patients in arm C.

DETAILED DESCRIPTION:
250 patients with locally advanced or metastatic gastric carcinoma or carcinoma of the esophagogastric junction without prior palliative therapy will be treated with 8 cycles of the FLOT scheme (up to 12 cycles if the response is favourable). Prior to enrolment a unique and detailed clinical evaluation of the dissemination of the disease will be done which includes a differentiated regard of the M-category in the TNM classification. A prospective stratification will classify the patients as having either (A) locally advanced, (B) limited metastatic, or (C) extensive metastatic disease. In addition, the pharmacogenetic risk profile of the patients will be evaluated by a combined analysis of two genetic polymorphisms of the metabolism of the applied substances (XPD312, GSTT1). For the assessment of the disease, reference regions are examined by CT or MRI scans and if applicable endoscopy prior to the start of the study, every 2 months during and after the end of therapy until progression of the disease occurs. Evaluation of quality of life (by standard forms like EORTC-Q30 and others) is continued after progression. Clinical examinations (blood count, assessment of toxicity, anamnesis) is performed every two weeks for evaluation of toxicity and application of chemotherapy. After informed consent is given, peripheral blood of the patient will be analysed for the pharmacogenetic risk profile. Representative tumor material will be analysed by immunohistochemistry and quantitative PCR for the expression of several molecular factors.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced gastric cancer or adenocarcinoma of the esophagogastric junction
* No prior chemotherapy in metastatic state
* Adequate blood and biochemistry parameters

Exclusion Criteria:

* Hypersensitivity for 5-FU, Leucovorin, Oxaliplatin or Docetaxel
* KHK, cardiomyopathy or cardiac insufficiency
* Malignancy <5 years ago
* Brain metastases
* Severe internal disease or inadequate blood and biochemistry parameters
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
overall survival | every 2 weeks during study, every 3 months follow-up

SECONDARY OUTCOMES:
Pharmacogenetic risk profile | once at beginning
Quality of Life | every 8 weeks
Progression free survival (PFS) and response rate (Stratum B and C) | every 8 weeks
rate of R0-resections, rate of pathological remissions and perioperative morbidity and mortality in stratum A and B Perioperative Morbidität und Mortalität in dem Arm A und ggf. B | after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batan, MD, Study Chair — Institute of Clinical Cancer Research IKF, UCT - University Cancer Center, Frankfurt, Germany
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany

REFERENCES:
- [Background] Al-Batran SE, Hartmann JT, Probst S, Schmalenberg H, Hollerbach S, Hofheinz R, Rethwisch V, Seipelt G, Homann N, Wilhelm G, Schuch G, Stoehlmacher J, Derigs HG, Hegewisch-Becker S, Grossmann J, Pauligk C, Atmaca A, Bokemeyer C, Knuth A, Jager E; Arbeitsgemeinschaft Internistische Onkologie. Phase III trial in metastatic gastroesophageal adenocarcinoma with fluorouracil, leucovorin plus either oxaliplatin or cisplatin: a study of the Arbeitsgemeinschaft Internistische Onkologie. J Clin Oncol. 2008 Mar 20;26(9):1435-42. doi: 10.1200/JCO.2007.13.9378. PMID 18349393
- [Background] Al-Batran SE, Hartmann JT, Hofheinz R, Homann N, Rethwisch V, Probst S, Stoehlmacher J, Clemens MR, Mahlberg R, Fritz M, Seipelt G, Sievert M, Pauligk C, Atmaca A, Jager E. Biweekly fluorouracil, leucovorin, oxaliplatin, and docetaxel (FLOT) for patients with metastatic adenocarcinoma of the stomach or esophagogastric junction: a phase II trial of the Arbeitsgemeinschaft Internistische Onkologie. Ann Oncol. 2008 Nov;19(11):1882-7. doi: 10.1093/annonc/mdn403. Epub 2008 Jul 31. PMID 18669868
- [Background] Al-Batran SE, Atmaca A, Hegewisch-Becker S, Jaeger D, Hahnfeld S, Rummel MJ, Seipelt G, Rost A, Orth J, Knuth A, Jaeger E. Phase II trial of biweekly infusional fluorouracil, folinic acid, and oxaliplatin in patients with advanced gastric cancer. J Clin Oncol. 2004 Feb 15;22(4):658-63. doi: 10.1200/JCO.2004.07.042. PMID 14966088
- [Derived] Al-Batran SE, Homann N, Pauligk C, Illerhaus G, Martens UM, Stoehlmacher J, Schmalenberg H, Luley KB, Prasnikar N, Egger M, Probst S, Messmann H, Moehler M, Fischbach W, Hartmann JT, Mayer F, Hoffkes HG, Koenigsmann M, Arnold D, Kraus TW, Grimm K, Berkhoff S, Post S, Jager E, Bechstein W, Ronellenfitsch U, Monig S, Hofheinz RD. Effect of Neoadjuvant Chemotherapy Followed by Surgical Resection on Survival in Patients With Limited Metastatic Gastric or Gastroesophageal Junction Cancer: The AIO-FLOT3 Trial. JAMA Oncol. 2017 Sep 1;3(9):1237-1244. doi: 10.1001/jamaoncol.2017.0515. PMID 28448662